CLINICAL TRIAL: NCT00366938
Title: A 13-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Trial of 2 Different Dose Regimens of Lumiracoxib (100 mg od and 200 mg od Initial Dose for Two Weeks Followed by 100 mg od) in Patients With Primary Knee Osteoarthritis, Using Celecoxib (200 mg od) as a Comparator
Brief Title: Efficacy and Safety of Lumiracoxib in Patients With Knee Osteoarthritis (OA).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2360
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, lumiracoxib, celecoxib, Cox-2
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study will investigate the efficacy and safety of lumiracoxib in patients with primary knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee (confirmed by American College of Rheumatology [ACR] criteria).
* Requirement of regular non-steroidal anti-inflammatory drug (NSAID) therapy.

Exclusion Criteria:

* Evidence of active gastrointestinal ulceration within 12 months prior to the screening visit or history of active gastrointestinal bleeding within the previous 5 years.
* Known hypersensitivity to analgesics, antipyretics, or NSAIDS (including celecoxib).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1464
Dates: Start 2003-09; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Overall OA pain intensity in the target knee using a 0-100 mm Visual Analogue Scale (VAS), at week 13.
Patient's global assessment of disease activity using a 0-100 mm VAS, at week 13.
Patient's functional status using Western Ontario and McMaster Universities Arthritis Index (WOMAC©) total score, at week 13.

SECONDARY OUTCOMES:
Overall OA pain intensity in the target knee using 0-100 mm VAS, at weeks 2, 4, 8.
Patient's global assessment of disease activity using 0-100 mm VAS, at weeks 2, 4, 8.
Patient's functional status using WOMAC© Likert 3.1 sub-scale scores and total score, at weeks 2, 8, 13.
Patient's health status using the Short Form-36 (SF-36), at week 13.
Physician's global assessment of disease activity using 0-100 mm VAS, at weeks 2, 4, 8.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis
Locations (1):
- Novartis Pharmaceuticals Corporation, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Dougados M, Moore A, Yu S, Gitton X. Evaluation of the patient acceptable symptom state in a pooled analysis of two multicentre, randomised, double-blind, placebo-controlled studies evaluating lumiracoxib and celecoxib in patients with osteoarthritis. Arthritis Res Ther. 2007;9(1):R11. doi: 10.1186/ar2118. PMID 17266764